CLINICAL TRIAL: NCT00392041
Title: Eszopiclone in the Treatment of Insomnia and Associated Symptoms of Fibromyalgia
Brief Title: Eszopiclone in the Treatment of Insomnia and Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lesley A. Allen, Ph.D. (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lesley A. Allen, Ph.D., Associate Professor of Psychiatry, University of Medicine and Dentistry of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0220060122
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Fibromyalgia; Insomnia
Keywords: Fibromyalgia; Insomnia; Sleep; Eszopiclone; Lunesta
MeSH Terms: conditions — Fibromyalgia; Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eszopiclone (Experimental)
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Eszopiclone — 3mg qpm for 12 weeks
  Other Names: Lunesta
  Arms: Eszopiclone
Drug: placebo — 1 pill qpm for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose is to assess the efficacy of eszopiclone for the treatment of insomnia and other symptoms of fibromyalgia. It is hypothesized that participants receiving eszopiclone will report greater improvement in total sleep time, sleep quality, pain, fatigue, physical functioning, and emotional distress than will those receiving placebo.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a prevalent, debilitating, and costly syndrome. Although the pathophysiology of FM is not yet well-understood, sleep disturbance is a prominent feature of most theories. Eszopiclone has been approved by the FDA for the treatment of insomnia, but has not been studied in the treatment of FMS. The purpose is to assess the efficacy of eszopiclone for the treatment of insomnia and other symptoms of fibromyalgia (FMS) in FMS patients. Participants will be randomly selected to receive eszopiclone or placebo. It is hypothesized that participants receiving eszopiclone will report greater improvement in total sleep time, sleep quality, pain, fatigue, physical functioning, and emotional distress than will those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 through 64.
2. Meets ACR criteria for FMS, as determined by rheumatological examination and a medical history review.
3. Reports sleep maintenance insomnia (total sleep time of < 6.5 hours or sleep impairment consisting of 3 of 7 nights per week for a month by history) or sleep onset latency insomnia (at least 3 of 7 nights of sleep latency > 30 minutes), as well as clinically significant daytime distress or impairment during the 1 week self assessment prior to baseline.
4. Has completed 8th grade and is fluent in English.
5. If a female of child bearing potential, the patient must be non-pregnant and either post-menopausal or using an approved birth control method. Acceptable birth control methods include: history of tubal ligation, having a male partner who is sterile, IUDs, birth control pills or other hormonal birth control methods (e.g., birth control patch, Depo-Provera injections), and double-barrier methods (e.g., condom and foam).
6. Antidepressant medication will be allowed if the patient has been on a stable dose for at least one month.

Exclusion Criteria:

1. Evidence of traumatic injury, inflammatory rheumatic disease, or infectious or endocrine-related arthropathy.
2. Evidence of a primary sleep disorder (e.g., significant sleep disordered breathing (central or obstructive apnea), periodic limb movement disorder, or REM sleep behavior disorder.
3. Any current, clinically significant medical condition.
4. Pregnancy.
5. Meets DSM-IV criteria for bipolar disorder, psychotic disorder, organic brain syndrome, or psychoactive substance abuse or dependence.
6. Any current psychiatric disorder that would interfere with study participation (investigator judgment).
7. Active suicidal ideation.
8. Plans to engage in additional psychotherapy during the study.
9. Concurrent use of benzodiazepines after 6pm or as a sleep aid.
10. Concurrent use of any other sleep aid.
11. Concurrent use of analgesics other than acetaminophen or non-steroidal anti-inflammatory medication.
12. Concurrent use of any medication that has not been stabilized for at least 1 month prior to screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley A. Allen, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Department of Psychiatry, UMDNJ-Robert Wood Johnson Medical School, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First 4 Weeks
Arm/Group | Eszopiclone | Placebo
Started | 19 | 17
Completed | 11 | 14
Not Completed | 8 | 3
Period: Weeks 5 - 12
Arm/Group | Eszopiclone | Placebo
Started | 11 | 14
Completed | 7 | 9
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone | Placebo | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.58 (8.60) | 46.94 (11.14) | 44.11 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Sleep Time (TST) as Recorded in Patient Diaries
Description: Difference in total sleep time between week 4 and baseline
Time Frame: week 4
Population: Data are reported through week 4, instead of through week 12 as planned, because of the high drop out rate after week 4. Fewer than 50% of participants remained in the study at week 12.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 19 | 17
minutes | 68.72 (69.72) | 13.47 (83.21)

2. Secondary Outcome: Wake Time After Sleep Onset (WASO)
Description: Minutes awake after sleep onset as recorded in patient diaries
Time Frame: week 12
Population: Data collected was of too poor quality to analyze in a meaningful way
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Sleep Quality
Time Frame: week 12
Population: Data recorded was of too poor quality to analyze in a meaningful way
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinician-rated Overall Severity of Fibromyalgia
Time Frame: week 12
Population: Data recorded was of too poor quality to analyze in a meaningful way
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Fibromyalgia Impact Questionnaire
Time Frame: week 12
Population: Data recorded was of too poor quality to analyze in a meaningful way
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No